CLINICAL TRIAL: NCT06013501
Title: The Effect of Puppet Show on Pain and Fear During Subcutaneous Injection in Children With Leukemia: A Randomized Controlled Study
Brief Title: The Effect of Puppet Show on Pain and Fear During Subcutaneous Injection in Children With Leukemia
Acronym: SC-puppet
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Collaborators: Ege University (Other)
Responsible Party: Principal Investigator, Gülçin Özalp Gerçeker, pHD, Assoc. Prof., Dokuz Eylul University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: SC-puppet
Record Dates: First submitted 2023-03-30; First posted 2023-08-28 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Pain, Acute; Fear
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Intervention Model Description: Randomised
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Puppet Show Group (Experimental): puppet show before and during subcutaneous injection
  Interventions: Behavioral: puppet show
- Control group (No Intervention): standart care

INTERVENTIONS:
Behavioral: puppet show — puppet show to the child before and during subcutaneous application
  Arms: Puppet Show Group

SUMMARY:
This study aim to evaluate the effect of puppet show applied during subcutaneous injection to children aged 3-7 years with leukemia on the level of pain and fear experienced by children due to the intervention.

DETAILED DESCRIPTION:
Before and during subcutaneous injection administration to the children in the study group There will be a puppet show. No distraction method will be applied to the children in the control group and the clinical A subcutaneous injection will be administered in accordance with the routine. Pain and fear assessment of children in both groups will be evaluated by the clinical nurse during the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Child <3 and >7 years old
* Medically unstable (dehydration, septic shock, sedation)
* Children who are being treated for leukemia in the Pediatric Hematology Service will be included in the study.

Exclusion Criteria:

* Not exposed to any other interventional procedure before (same day) subcutaneous intervention
* Not expressing any pain before subcutaneous intervention
* Heart rate to be within age-appropriate limits
* Wong-Baker Pain Rating Scale score of 0 in the evaluation performed before the subcutaneous intervention (5 minutes ago)
* Having a disability that cannot perceive the attempt and communicate (down syndrome, speech disorder, visual impairment)
* The child and family do not know Turkish

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2023-01-03 (Actual); Primary Completion 2024-12-03 (Estimated); Study Completion 2024-12-03 (Estimated)

PRIMARY OUTCOMES:
procedure-related pain with Wong Baker Pain Rating Scale | change from Wong Baker Pain Rating Scale (5 minutes before the subcutaneous injection, 5 minutes after subcutaneous injection)
  pain assessment with Wong Baker Pain Rating Scale by child
procedure-related fear with Child Fear Scale | change from Child Fear Scale (5 minutes before the subcutaneous injection, 5 minutes after subcutaneous injection)
  fear assessment with Child Fear Scale by child and parent
procedure-related pain with The FLACC scale or Face, Legs, Activity, Cry, Consolability scale | change from The FLACC scale or Face, Legs, Activity, Cry, Consolability scale (5 minutes before the subcutaneous injection, 5 minutes after subcutaneous injection)
  pain assessment with The FLACC scale or Face, Legs, Activity, Cry, Consolability scale by nurse

SECONDARY OUTCOMES:
Heart rate | change from the heart rate at 10 minutes
  Heart rate measurement

CONTACTS AND LOCATIONS:
Overall Officials: Gülçin Özalp Gerçeker, pHD, Principal Investigator — Dokuz Eylul University
Locations (1):
- Gülçin Özalp Gerçeker, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No